CLINICAL TRIAL: NCT01045616
Title: Evaluation of Refractive Status and Ophthalmological Problems of Prematurity
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: CHUNG-MAY YANG, MD, Department of Ophthalmology, National Taiwan University Hospital
Other Study IDs: 200806070R
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prematurity

SUMMARY:
Children born with very low birth weight and extremely low birth weight are at increased risk of various ophthalmic challenges such as retinopathy of prematurity (ROP), refractive error, strabismus, cerebral visual impairment, colour vision deficits, reduced contrast sensitivity (CS), visual field defects, and decreased visual acuity (VA). Many of these factors are not independent of each other. Among them, refractive error is a really common disorder. These can cause significant disability which can impact life's activities and, qualities. Currently, no standard guidelines are available toward the provision of ophthalmic follow up care for preterm infants. It is important to survey the prevalence of different ophthalmic sequelae in Taiwan, to identify the risk factors of developing these sequelae, and, furthermore, to build up a screening program. The preterm population has heterogeneous conditions to developing ophthalmic sequelae. National Taiwan University Hospital (NTUH) is now in charge of a big part of intense care for these low birth weight preterm neonates. With detailed medical record done of these children during care in the neonatal unit, we are competence for this meaningful program.

DETAILED DESCRIPTION:
Improved neonatal care has resulted in the reduced mortality of preterm infants, especially in the very low birth weight and extremely low birth weight groups. However, this reduced mortality can be associated with long-term medical sequelae. For example, preterm infants are at increased risk of chronic illnesses such as cerebral palsy and asthma, as well as having poor motor skills, poor adaptive functioning, and low intelligence quotient.

As for the ophthalmic problems, ophthalmic challenges following preterm birth are numerous and morbid ocular conditions are not rare. The threat to visual development of prematurity does not end when the retina is fully vascularised and the risk of ROP has passed. The risk of blindness for babies of birth weight <1500 g is increased over 25 times compared to children born at full term. The conditions which result severe visual loss include ROP, cerebral vision impairment, cataracts and optic atrophy, whereas other conditions, primarily amblyopia, may result in better visual outcome. Effects of prematurity on ocular and neurological development include retinopathy of prematurity (ROP), refractive error, strabismus, cerebral visual impairment, colour vision deficits, reduced contrast sensitivity (CS), visual field defects, and decreased visual acuity (VA). Many of these factors are not independent of each other. Among them, refractive error is a really common disorder. These can cause significant disability which can impact life's activities and, qualities.

There are numerous reports of an increase refractive errors and amblyogenic factors in the low birth weight population relative to children born at full term. However, no formal database was established in Taiwan. Today in Taiwan, with increasing level of educational and living standard, the prevalence and severity of myopia and other refractive errors appear to be an upward trend. The rate is much higher than other developed countries and both genetic and environmental factors are crucial to it. Under such as a special condition, the tendency of increasing refractive errors and amblyogenic factors in the low birth weight children is questionable and need our effort to identify them.

Currently, no standard guidelines are available toward the provision of ophthalmic follow up care for preterm infants. For most preterm children born in Taiwan, between the time of discharge from the neonatal unit until national screening at 6-7 years of age (receiving education in elementary school), there is no routine ophthalmic surveillance. Due to the concern of life's activities and qualities of these children, it is important to survey the prevalence of different ophthalmic sequelae in Taiwan, to identify the risk factors of developing these sequelae, and, furthermore, to build up a screening program. The preterm population has heterogeneous conditions to developing ophthalmic sequelae. To use limited health service resources efficiently, it would be helpful to identify those who are at high risk of developing ophthalmic sequelae. National Taiwan University Hospital (NTUH), as one of the largest tertiary medical centers in northern Taiwan, is now in charge of a big part of intense care for these low birth weight preterm neonates. With detailed medical record done of these children during care in the neonatal unit, we are competence for this meaningful program.

ELIGIBILITY:
Inclusion Criteria:

* (1) born at post-conception age of less than 35 weeks or with birth weight of less than 1500 gm.
* (2) complete medical records and ophthalmic records available

Exclusion Criteria:

* if unable to communicate or have ophthalmological examinations done due to cognitive defect.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with premature birth history born between January 1, 1999 and December 30, 2001 in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The refractive status of these children born prematurely | from 2008/7 - 2009/12

SECONDARY OUTCOMES:
other ophthalmological problems of these children born prematurely | from 2008-7 to 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: CHUNG-MAY YANG, MD, Study Director — National Taiwan University Hospital; Tzu-Hsun Tsai, MD, Study Director — National Taiwan University Hospital; Ta-Ching Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen TC, Tsai TH, Shih YF, Yeh PT, Yang CH, Hu FC, Lin LL, Yang CM. Long-term evaluation of refractive status and optical components in eyes of children born prematurely. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6140-8. doi: 10.1167/iovs.10-5234. Epub 2010 Aug 4. PMID 20688740